CLINICAL TRIAL: NCT04384640
Title: The Effect of Patient's Position After Intra-tympanic Injection on the Amount of Fluid in the Middle Ear
Brief Title: The Effect of Patient's Position After Intra-tympanic Injection
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0182-20-TLVMC
Record Dates: First submitted 2020-05-08; First posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Sudden Hearing Loss
MeSH Terms: conditions — Hearing Loss, Sudden

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients seated after Intra-Tympanic injection
  Interventions: Other: Change of posture after Intra Tympanic injection

INTERVENTIONS:
Other: Change of posture after Intra Tympanic injection — Seating position after Intra Tympanic injection

SUMMARY:
The effect of the patient's head on the leakage of steroids from the middle ear to the throat will be studied. The patients will be seated after one of the intra tympanic injections that are routonely performed due to Sudden Sensorineural Hearin Loss (SNHL). The patients will be asked if they taste the steroids in their throats.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Sudden Sensorineural Hearing Loss, treated using intra-tympanic injection of steroids
* Patients who signed an informed consent form

Exclusion Criteria:

* Dysgeusia
* Inner or middle ear malfomation
* Eustachian tube dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Sudden Sensorineural Hearing Loss, treated using intra-tympanic injection of steroids
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Degree of taste | 0 Minutes, and then 10, 20, 30 minutes after the injection
  The patients will rate the degree of change of taste in their throat

IPD SHARING:
Plan to Share IPD: No